CLINICAL TRIAL: NCT00251537
Title: A Pilot Study Assessing Safety and Antiretroviral Activity of Intravenously Administered LTB4 in HIV-1 Infected Adults With a CD4 Count Greater Than 250 Cells/mm3 and a Viral Load Greater Than 5,000 Copies/mL, and Who Have Not Received Antiretroviral Therapy Within Two Months
Brief Title: A Pilot Study of LTB4 in HIV-1 Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LTB4 Sweden AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTB4 200501
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: Pilot study; Randomized; Placebo-controlled; Double-blind; Effect on viral load; LTB4; HIV-1 infection
MeSH Terms: conditions — HIV Infections | interventions — Leukotriene B4

INTERVENTIONS:
Drug: LTB4

SUMMARY:
This is a pilot study to assess the safety and antiretroviral activity of a naturally occuring substance known as Leukotriene B4(LTB4). The aim of the study is to determine the effect of LTB4 on viral load during a period of 6 weeks, 4 weeks of active treatment and 2 additional weeks after the end of active treatment for safety follow-up. 40 patients in seven clinics in Canada will be randomized into three treatment arms, either of two doses of LTB4 or placebo. Study drug is administered intravenously once daily. LTB4 can activate and stimulate various white blood cells and by the activation release natural substances in the body and this process is an important part of the body's defense against infections.

DETAILED DESCRIPTION:
The objective of this pilot study is to investigate whether LTB4, administered at a dose that provides an increase in alfa-defensin release from neutrophils, can affect HIV viral load in HIV-1 infected individuals. The safety, tolerability and effect will be assessed of 28 days of daily intravenous dosing of LTB4 on HIV viral load. Safety and tolerability will also be assessed.

The study is randomized, double-blind, placebo controlled. All subjects will be randomly assigned to one of three treamtent groups, LTB4 at two different dose levels or corresponding placebo. Treatment duration is 4 weeks and follow-up period is 2 weeks. Subjects will visit the clinic on a daily basis during the treatment period to receive a daily intravenous injection of the study drug. 40 subjects will be enrolled, seven clinics in Canada will participate in the study.

Primary endpoint: Change in viral load over the treatment period of 28 days. Secondary endpoint: CD4, CD8 and neutrophil counts, alfa-defensins and CC-che, mokine release in blood.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 18 and 65 years of age
2. Diagnosis of HIV-1 infection
3. Plasma HIV RNA level greater or equal to 5,000 copies/mL at the screening visit
4. A CD4 cell count equal or greater than 250 cells/mm3 and CD4 fraction equal or greater than 14% at the screening visit within one month of study entry
5. No ART within two months of study entry
6. Karnofsky score equal to or above 80
7. If female of childbearing potential, a negative serum pregnancy test at screening.
8. In the opinion of the investigator, the subject will be able to comply with the requirements of the protocol, including ability to present for all required visits
9. Subject is capable of understanding and signing an informed consent form

Exclusion criteria:

1. Primary HIV-1 infection
2. Use of investigational therapy in the preceding month prior to screening visit
3. Prior screening for entry into this study
4. Use of G-CSF, GM-CSF, IL-2, IFNs, erythropoietin, systemic or inhaled steroids within one month of the screening visit
5. HIV-vaccine within one year of the screening visit
6. Concurrent disease or conditions that may present a risk to the subjects
7. Females who are pregnant or breast feeding
8. History of any malignancy or any active malignancy, except cutaneous Kaposis sarcoma
9. Unexplained temperature of 38.5 degrees Celsius
10. Chronic diarrhea (>3 liquid stools per day persisting for 15 days) within one month prior to study entry
11. Calculated creatinine clearance outside normal limits
12. Urinalysis: hemoglobinuria, present
13. Liver transaminases > 3 x ULN
14. Absolute neutrophil count < 500/mm3
15. Hemoglobin < 8.0g/dL
16. Platelet count < 75,000/mm3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-11; Study Completion 2006-08

PRIMARY OUTCOMES:
To assess the effect of 28 days of daily dosing of LTB4 on HIV viral load

SECONDARY OUTCOMES:
To assess safety and tolerability of 28 days of daily dosing
To assess effects on CD4 and CD8 counts of 28 days of daily dosing
To assess effects on neutrophil counts of 28 days of dosing
To assess effects on release of alfa-defensins and CC-chemokines in blood on day s 1, 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lalonde, MD, Principal Investigator — Montreal Chest Institute, Montreal, Canada
Locations (7):
- Canada (7):
  - Centre for HIV/AIDS, St Pauls Hospital, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - The Ottawa Hospital (General Campus), Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec